CLINICAL TRIAL: NCT06150859
Title: Efficacy of Ayahuasca in Concert With Psychotherapy to Decrease the Severity of Grief
Brief Title: Ayahuasca Assisted Psychotherapy for Grief
Acronym: PSICODUELAYA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Beckley Med Foundation (Other)
Responsible Party: Principal Investigator, Débora González, Principal Investigator, Beckley Med Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI-19-118
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Bereavement
Keywords: Bereavement; Ayahuasca; Psychotherapy; Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Ayahuasca-assisted constructivist therapy. (Experimental): Constructivist psychotherapy will be delivered over 9 online psychotherapeutic sessions interconnected in 3 modules to process trauma, restore attachment security and reconstruct the self. One preparation session and two integration sessions after two ayahuasca administrations are included to the experimental group.
  Interventions: Drug: Ayahausca-Assisted psychotherapy
- Constructivist Psychotherapy (Active Comparator): Constructivist Psychotherapy will be delivered over 9 online psychotherapeutic sessions interconnected in 3 modules to process trauma, restore attachment security and reconstruct the self.
  Once the follow-up period is over (3 months), participants have the option of receiving 2 administrations of ayahuasca if the severity of grief is high.
  Interventions: Behavioral: Constructivist Psychotherapy
- No treatment (Other): Participants received no treatment during the 9-week Control Period.
  Once the follow-up period is over (3 months), participants have the option of receiving 2 administrations of ayahuasca if the severity of grief is high.
  Interventions: Other: No treatment

INTERVENTIONS:
Drug: Ayahausca-Assisted psychotherapy — Drug: Two ayahuasca administrations (0.75 mg/kg DMT), after 3rd and 6th therapeutic session. Ayahuasca is a psychoactive mixture of plants which contains DMT as an active principle.
  Constructivist Psychotherapy will be delivered over 9 online psychotherapeutic sessions.
  Other Names: Ayahausca-assisted grief therapy
  Arms: Experimental: Ayahuasca-assisted constructivist therapy.
Behavioral: Constructivist Psychotherapy — Constructivist Psychotherapy will be delivered over 9 online psychotherapeutic sessions
  Arms: Constructivist Psychotherapy
Other: No treatment — No treatment during the control period
  Arms: No treatment

SUMMARY:
The aim of this study is to compare the effectiveness of an ayahuasca-assisted constructivist therapy with constructivist therapy and no treatment to decrease the severity of grief. A secondary purpose is to assess the effectiveness to prevent Persistent Complex Bereavement Disorder and Prolonged Grief Disorder, and to assess potential changes in avoidance, meaning-making and self-clarity. Subjective effects and Acceptance promoting effects of psychedelic drug are assessed after ayahuasca administration. A non-randomized controlled trial is proposed with three arms involving an experimental group (ayahuasca in concert with psychotherapy) and two control groups (psychotherapy and no treatment) with pretest, posttest and 3 months follow-up.

DETAILED DESCRIPTION:
Grief is a deep and intense sorrow caused by the loss of someone loved. Although every person could benefit from support, only a substantial minority of bereaved people experience severe, persistent and disabling grief (PCBD), requiring treatment one year after the death of a loved one. However, pharmacotherapy alone has not proven to be effective, and while psychological interventions for prolonged grief disorder may be efficacious, the clinical effectiveness is small (Hedges' g: 0.41-0.45). As far as we know, no bereavement prevention program has proven to be effective, and early interventions are discouraged. Thus, there are no effective resources for supporting the bereaved during the months following the death of a loved one, a need which peaks during the months following the death, when grief is most intense and the bereaved lives are at their highest level of risk.

ELIGIBILITY:
Inclusion Criteria:

* Experienced the loss of a first- degree relative not more than 12 months prior to enrollment as indicated by self-report.
* Scores up to 40 in the Texas Revised Inventory of Grief (TRIG).

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Hypertension (systolic blood pressure above 140 mm, diastolic above 90 mm and heart rate above 100 bpm).
* History of psychotic disorder (Axis I-II of the DSM-V).
* Substance use disorder (except nicotine).
* Alcohol consumption greater than 40 g/day.
* Receiving psychological or self-help therapy during the study on a regular basis.
* Receiving regular pharmacological therapy for complicated grief during the study.
* Regular intake of any type of medication in the month preceding the study.
* Treatment with single doses of symptomatic medication during the study may be accepted (as long as it can be assumed that the ingested drug has been completely eliminated on the days of the ayahuasca administrations).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in the severity of grief symptoms | Time Frame: Baseline to End of Intervention, up to 3 months
  Change in grief severity is measured by the present scale of Texas- Revised Grief Inventory (TRIG), a measure of normal grief symptoms. For the TRIG the minimum units are 0 and Maximum units on the total scale are 65. The higher the number on the TRIG, the more severe the symptoms.

SECONDARY OUTCOMES:
Prevalence of Persisten Complex Bereavement (PCBD) and prolonged Grief Symptoms (PGD). | Baseline to End of Intervention, up to 3 months
  Measured using the Traumatic Grief Inventory self-report version (TGI-SR). The TGI-SR is a 18-item self-report measure to assess symptoms of Persistent Complex Bereavement Disorder (PCBD) included in Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 and Prolonged Grief Disorder (PGD). A score of ≥61 optimally classified participants as meeting criteria for PCBD-caseness and a score of ≥59 classified participants as meeting criteria for PGD-caseness.

OTHER OUTCOMES:
Individual's quality of life | Baseline to End of Intervention, up to 3 months
  Measured using the World Health Organization Quality of Life-Bref (WHO-qol-BREF). The WHO-qol-BREF has 26 items rated on 4 answer options. Only subscales on physical health, pshychological health and social relationships were included in this study. Higher scores indicate a better subjective QOL.
Posttraumatic Growth | Baseline to End of Intervention, up to 3 months
  Measured using the Posttraumatic Growth Inventory Short-Form (PSI-SF). The PSI-SF has 10 items rated on 6-point Likert scale ranging from 1 ("completely disagree") to 6 ("completely agree"). This questionnaire includes 4 sub scales: New Possibilities, Personal Strength, Spiritual Change, and Appreciation of Life. Higher scores indicate a higher posttraumatic growth.
Avoidance | Measured using the Acceptance and Action Questionnaire (AAQ-II). The AAQ-II has 7 items rated on a 7-point Likert scale ranging from 1 ("never true") to 7 ("always true") to assess indirectly acceptance. Higher scores indicate a higher avoidance.
  Baseline to End of Intervention, up to 3 months
Meaning-made | Baseline to End of Intervention, up to 3 months
  Measured using the Stressful Life Experiences Scale (ISLES-SF). The ISLES-SF has 6 items rated on a 5-point Likert scale, ranging from 1 ("completely agree") to 5 ("completely disagree"). The questionnaire includes two subscales: Comprehensibility and Footing in the World. Higher scores indicate more adaptive meaning made of a loss.
  Baseline to End of Intervention, up to 3 months
Consistency of self beliefs | Baseline to End of Intervention, up to 3 months
  Measured using the Self-concept Clarity Scale (SCS). The SCS has 12 items rated on a 7-point Likert scale ranging from 1 ("strongly disagree") to 7 ("strongly agree"). Higher scores reflect greater self-concept clarity.
Subjective effects of ayahuasca. | 3 days after each ayahuasca administration
  Measured using the Five Dimensional Altered States of Consciousness" (5D-ASC). The 5D-ASC has items rated on a 100-point Likert scale ranging from 0 ("No, no more than usually) to 100 ("Yes, much more than usually"). The questionnaire includes three subscales: Visionary Restructuralization, Oceanic Boundlessness and Anxious Ego-Dissolution
Acceptance promoting effects of psychedelic drug | 3 days after each ayahuasca administration
  Measured using the Acceptance/Avoidance-Promoting Experiences Questionnaire (APEQ). The APEC has 32 items rated on a 0 ("No, not at all") and 100 ("Yes, extremely or absolutely"). The questionnaire includes two main scales, acceptance-related experience (ACE) and avoidance-related experience (AVE).

CONTACTS AND LOCATIONS:
Overall Officials: Magi Farré, Study Director — Hospital German Trials I Pujol
Locations (1):
- Institut de Recerca Holistica de Montserat (Irehom), Barcelona, Spain

REFERENCES:
- [Derived] Sabucedo P, Andion O, Neimeyer RA, Soto-Angona O, Javkin J, Haro JM, Farre M, Gonzalez D. Ayahuasca-assisted meaning reconstruction therapy for grief: a non-randomized clinical trial protocol. Front Psychiatry. 2025 Jan 7;15:1484736. doi: 10.3389/fpsyt.2024.1484736. eCollection 2024. PMID 39839135